CLINICAL TRIAL: NCT00149474
Title: Peak Flow Monitoring in Older Adults With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized
Other Study IDs: 260; R01HL052598 (NIH)
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2005-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Behavioral: Peak Flow Monitoring

SUMMARY:
Evaluate the incremental effectiveness of peak flow monitoring ove symptom monitoring as a management tool to enhance asthma control in adults >= 50 years with moderate-severe asthma.

DETAILED DESCRIPTION:
BACKGROUND:

We propose a five-year Demonstration and Education project to assess the incremental value of peak flow monitoring (PFM) over symptom monitoring (SM) as a management tool for asthma control in adults greater than or equal to 50 years with moderate-severe asthma. We will develop three parallel asthma education programs for older adults using as our base an existing asthma education program (AIR/Kaiser Adult Education Program) of demonstrated efficacy for adults ,50 years of age.

DESIGN NARRATIVE:

Primary outcome Frequency and cost of health care utilization for asthma, and asthma-specific quality of life

Key secondary outcomes Prebronchodilator FEV1; diurnal variability in PEF

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Inclusions: Doctor-diagnosed asthma; >=50 years; using asthma medications; >12% increase in FEV1 after two puffs of inhaled beta-agonist; willing to participate in asthma meducation program and two-year follow up; likely to stay in Portland area; KPNW member for two years.

Exclusions: Unable to read, speak or understand English; no telephone; failure to keep two pre-randomization appointments; inability to reproducible FEV 1 maneuver; participation in pilot phase of study; concurrent participation in any other medical research study.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1994-08; Study Completion 1999-07 (Actual)